CLINICAL TRIAL: NCT05057182
Title: mRNA Vaccination to Boost Antibodies Against SARS-CoV-2 in Recipients of Inactivated Vaccines (the "mBoost" Study)
Brief Title: Third Dose of mRNA Vaccination to Boost COVID-19 Immunity (mBoost Study)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BJC050
Record Dates: First submitted 2021-09-24; First posted 2021-09-27 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: COVID 19 Vaccine
MeSH Terms: interventions — BNT162 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BNT162b2 (Experimental): BNT162b2 mRNA vaccine (Cominarty®, BioNTech/Fosun Pharma), one dose (0.3mL after dilution) contains 30 micrograms of COVID-19 mRNA Vaccine embedded in lipid nanoparticles.
  Interventions: Biological: BNT162b2

INTERVENTIONS:
Biological: BNT162b2 — BNT162b2 mRNA vaccine (Cominarty®, BioNTech/Fosun Pharma), one dose (0.3mL after dilution) contains 30 micrograms of COVID-19 mRNA Vaccine embedded in lipid nanoparticles.
  Other Names: Comirnaty

SUMMARY:
300 adults ≥30 years of age who have previously received two doses of an inactivated COVID-19 vaccine at least 3 months earlier will receive a third dose with an mRNA vaccine (BNT162b2, BioNTech). Investigators will monitor reactogenicity and measure the immune response to the third dose.

DETAILED DESCRIPTION:
Background: The accrual of population immunity to COVID-19 could allow life to return to pre- pandemic normality. Immunity can be acquired through natural infections or, preferably, by vaccination. An unprecedented global effort has succeeded in developing a number of COVID-19 vaccines. All vaccines against COVID-19 approved until now have originally been developed as either a single dose or following a homologous two-dose regimen. Inactivated COVID-19 vaccines have shown inferior immunogenicity compared to mRNA vaccines but there are no studies looking into the immunogenicity, reactogenicity and safety profile of mRNA vaccination provided as a booster dose in individuals who have previously received two doses of an inactivated COVID-19 vaccine.

Aims and Objectives: The aims of this study are: (1) to determine whether one dose of mRNA vaccine can boost neutralizing antibodies against SARS-CoV-2 in individuals who have previously received two doses of inactivated COVID-19 vaccines, and (2) to assess the reactogenicity and safety of heterologous 3rd doses of vaccination. The specific primary objective of this study is to assess the vaccine (humoral) immunogenicity, proxy by SARS-CoV-2 serum neutralizing antibody titers, of a 3rd dose dose of mRNA vaccine (using BNT162b2, Fosun/BioNTech) at 28 days after the booster dose in individuals who have previously received two doses of any inactivated COVID-19 vaccines.

Study design: Open label trial in adults aged 30 years of age or older (at enrolment). The duration of participation for each participant will be 12 months from the administration of the 3rd vaccine dose. The immune response and reactogenicity of one dose of BNT162b2 will be investigated in individuals who previously received two doses of any inactivated COVID-19 vaccines at least 3 months earlier. Participants will be enrolled shortly before receiving the booster dose of BNT162b2 (day 0), with blood collection at days 0, 28, 182 and 365 days after enrolment for analysis of humoral immune responses.

Main outcomes: The primary outcome is the vaccine immunogenicity measured as SARS-CoV-2 serum neutralizing antibodies in individuals who previously received two doses of any inactivated COVID-19 vaccines, evaluated as the geometric mean titer (GMT) at 28 days after the 3rd dose. The secondary outcomes include (1) a comparison of SARS- CoV-2 serum neutralizing antibodies as the geometric mean fold rise from baseline to each post-vaccination timepoint (i.e. at days 28, 182 and 365), and (2) descriptive analysis of the reactogenicity and safety profile of the 3rd dose.

Target population: Adults aged 30 years or older

Number of Subjects Planned: 300 participants to be recruited between September 2021 and December 2021

Study duration: 12 months for each participant

Potential implications: This study will provide important evidence into the effects of using a 3rd dose of mRNA vaccines to boost the immune response in individuals that had previously received two doses of inactivated vaccines. This information together with data collected on reactogenicity and safety could inform COVID-19 vaccination policy locally and internationally.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30 years or older at enrolment.
* Have received two doses of any inactivated COVID-19 vaccines (for example Sinovac- CoronaVac, Sinopharm-BIBP) with the most recent dose at least 90 days prior to enrolment.
* Currently resident and planning to remain resident in Hong Kong during the duration of the study, i.e. for 12 months after enrolment.
* Agreement to refrain from blood donation during the course of the study.
* Willing to provide blood samples for all the required time points.
* The individual or their caregiver have a home phone or cellular or mobile phone for communications purpose.
* Capable of providing informed consent.

Exclusion Criteria:

* A history of laboratory-confirmed or clinically confirmed COVID-19 infection. Have received (at least one dose of) any COVID-19 vaccines other than inactivated vaccines.
* Individuals who report any medical condition, or as determined by a clinician, not suitable to receive mRNA vaccines, including but not limited to allergies to the active substance or other ingredients of the vaccine.
* With diagnosed medical conditions related to their immune system.
* Use of medication that impairs immune system in the last 6 months, except topical steroids or short-term oral steroids (course lasting ≤ 14 days).
* Have used immunoglobulins and/or any blood products within 90 days prior to enrolment (administration of the study vaccine).
* Pregnancy, lactation or intention to become pregnant in the coming 3 months.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Titer of SARS-CoV-2 serum neutralizing antibodies | 28 days after vaccination
  The primary outcome measure is the vaccine (humoral) immunogenicity at 28 days after the booster dose of BNT162b2 in individuals who have previously received two doses of any inactivated COVID-19 vaccines, measured as geometric mean titer (GMT) of SARS-CoV-2 serum neutralizing antibodies using plaque reduction neutralization test (PRNT).

SECONDARY OUTCOMES:
Geometric Mean Titer of SARS-CoV-2 serum neutralizing antibodies | 182 and 365 days after vaccination
The geometric mean fold rise (GMFR) of SARS-CoV-2 serum neutralizing antibody titers from baseline to each post-vaccination timepoint measured. | Day 28, 49, 182 and 365 after vaccination
Reactogenicity | 7 days after vaccination or until the last symptom disappears
  Incidence of solicited local and systemic adverse events after the booster dose of vaccination.
Hospitalizations from any cause | 365 days after vaccination
  Incidence of hospitalizations during the year after receipt of the booster dose.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Cowling, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Shiu EYC, Cheng SMS, Martin-Sanchez M, Au NYM, Chan KCK, Li JKC, Fung LWC, Luk LLH, Chaothai S, Kwan TC, Ip DKM, Leung GM, Poon LLM, Peiris JSM, Leung NHL, Cowling BJ. Durability for 12 months of antibody response to a booster dose of monovalent BNT162b2 in adults who had initially received 2 doses of inactivated vaccine. Vaccine. 2024 Dec 2;42(26):126317. doi: 10.1016/j.vaccine.2024.126317. Epub 2024 Sep 13. PMID 39276621
- [Derived] Leung NHL, Cheng SMS, Martin-Sanchez M, Au NYM, Ng YY, Luk LLH, Chan KCK, Li JKC, Leung YWY, Tsang LCH, Chaothai S, Kwan KKH, Ip DKM, Poon LLM, Leung GM, Peiris JSM, Cowling BJ. Immunogenicity of a Third Dose of BNT162b2 to Ancestral Severe Acute Respiratory Syndrome Coronavirus 2 and the Omicron Variant in Adults Who Received 2 Doses of Inactivated Vaccine. Clin Infect Dis. 2023 Feb 8;76(3):e299-e307. doi: 10.1093/cid/ciac458. PMID 35675370